CLINICAL TRIAL: NCT04352114
Title: A Single-Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of LY3461767 in Healthy Participants
Brief Title: A Study of LY3461767 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 17517; J2L-MC-EZBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-04-16; First posted 2020-04-20 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY3461767 - Subcutaneous (SC) (Experimental): LY3461767 administered SC.
  Interventions: Drug: LY3461767 - SC
- Placebo - SC (Placebo Comparator): Placebo administered SC.
  Interventions: Drug: Placebo - SC
- LY3461767 - Intravenous (IV) (Experimental): LY3461767 administered IV.
  Interventions: Drug: LY3461767 - IV

INTERVENTIONS:
Drug: LY3461767 - SC — Administered SC.
  Arms: LY3461767 - Subcutaneous (SC)
Drug: LY3461767 - IV — Administered IV.
  Arms: LY3461767 - Intravenous (IV)
Drug: Placebo - SC — Administered SC.
  Arms: Placebo - SC

SUMMARY:
The main purpose of this study in healthy participants is to learn more about the safety of LY3461767 and any side effects that might be associated with it. The study will also measure how much LY3461767 gets into the bloodstream and how long it takes the body to get rid of it. For each participant, the study will last about 11 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Are healthy males, or females of non-child-bearing potential
* Have a body mass index of 18 to 35 kilograms per square meter (kg/m²)
* Have clinical laboratory tests within normal ranges as judged by investigator
* Have pulse rate and blood pressure within normal ranges as judged by investigator

Exclusion Criteria:

* Have Troponin I results above the upper reference limit, and judged to be clinically significant by the investigator, at screening
* Have an abnormality in the 12-lead electrocardiogram (ECG) at screening
* Have a significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal (GI), endocrine, hematological, or neurological disorders
* Regularly use known drugs of abuse
* Have donated blood of more than 450 milliliters (mL), or have participated in a clinical study that required similar blood volume collected within the past 3 months
* Have an average weekly alcohol intake that exceeds 7 units per week or are unwilling to stop alcohol consumption as required during the study
* Smoke more than 10 cigarettes per day
* Are current or former smokers with 30-pack-year smoking history
* Have a diagnosis or history of any malignancy
* Have not had appropriate cancer screening, in accordance with country specific guidance

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Day 29
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of LY3461767 | Baseline through Day 29
  PK: Cmax of LY3461767
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3461767 | Baseline through Day 29
  PK: AUC of LY3461767

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (2):
  - Covance Clinical Research Inc, Daytona Beach, Florida
  - Covance Dallas, Dallas, Texas
- Lilly Nus Centre for Clin Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No